CLINICAL TRIAL: NCT04242849
Title: IDH1/2 Mutational Analysis in AML Patients: Diagnosis and Follow-up
Status: Completed | Type: Observational
Sponsor: Josep Carreras Leukaemia Research Institute (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: N/A-NI-AML-PI-007344
Record Dates: First submitted 2020-01-16; First posted 2020-01-27 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2020-01

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Samples of bone marrow and peripheral blood of patients with AML
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- IDH1/2 mutated patients: Patients harboring mutations in IDH1 or IDH2 genes
- Patients without IDH1/2 mutations: Patients that don´t present any mutation in IDH1/2 genes

SUMMARY:
In a spanish series of AML patients it is intended to perform, at the moment of diagnosis, pyrosequencing of IDH1 and IDH2 genes. Taking into account the incidence of AML in the area, it is planed to study 100 patients per year.

Among the cases with IDH1/2 mutations, targeted deep sequencing (TDS) of a panel covering coding regions of 40 myeloid related genes will be applied. With TDS, pyrosequencing results will be validated at the same time that prognosis value of co-mutated genes could be studied. Furthermore, with TDS, molecular architecture of IDH1 and IDH2 mutated cases might be better understood.

ELIGIBILITY:
Inclusion Criteria:

* Patients >18 years old with de novo acute myeloid leukemia will be included. All patients will be treated according to clinical routine.

Exclusion Criteria:

* Patients not following the above criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients >18 years old with de novo acute myeloid leukemia (AML).
Sampling Method: Non-Probability Sample
Enrollment: 354 (Actual)
Dates: Start 2016-05-23 (Actual); Primary Completion 2019-12-27 (Actual); Study Completion 2020-01-16 (Actual)

PRIMARY OUTCOMES:
Presence of IDH1/2 mutation | 1 day
  Detection of mutations in IDH1 and IDH2 genes

SECONDARY OUTCOMES:
Detection of co-mutations | 1 day
  Screening of aditional mutations in those cases with IDH1/2 mutation

IPD SHARING:
Plan to Share IPD: No